CLINICAL TRIAL: NCT04633876
Title: Effects of 10 Weeks of Lifestyle Coaching on Cardiometabolic Risk Factors, Workability and Subjective Wellbeing - A Randomized Controlled Study
Brief Title: Effects of 10 Weeks of Lifestyle Coaching on Cardiometabolic Risk Factors, Workability and Subjective Wellbeing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Aava Medical (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); Finnish Institute of Occupational Health (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Virta1
Record Dates: First submitted 2020-05-19; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Work Related Stress; Metabolic Syndrome; Lipid Metabolism Disorders; Lifestyle Risk Reduction; Burnout
MeSH Terms: conditions — Occupational Stress; Metabolic Syndrome; Lipid Metabolism Disorders; Risk Reduction Behavior; Burnout, Psychological | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: RCT, lifestyle coaching in two arms: individualised coaching and group coaching. No coaching as a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): The subjects allocated to this group receive some results from baseline measurements (as do subjects in the intervention) but do not receive lifestyle counselling
  Interventions: Other: Control group
- Individual coaching (Experimental): These subjects receive individual counselling during the study.
  Interventions: Behavioral: Individual coaching
- Group coaching (Experimental): These subjects receive individual counselling during the study.
  Interventions: Behavioral: Group coaching

INTERVENTIONS:
Behavioral: Individual coaching — Individual coaching on lifestyle change, sleep, nutrition, physical activity and stress management.
  Arms: Individual coaching
Behavioral: Group coaching — Group coaching on lifestyle change, sleep, nutrition, physical activity and stress management.
  Arms: Group coaching
Other: Control group — Group receives no lifestyle coaching but did get baseline results from assessments which might motivate for lifestyle change.
  Arms: Control group

SUMMARY:
The main purpose of this study is to understand the impact of lifestyle coaching on the risk of future cardiometabolic disease, workability and self-assessed wellbeing. The data gathered during the study helps in the future to better identify different focus groups for more tailored interventions.

The study consists of two main stages: screening and coaching phase. Screening Aava and the pension will recruit 2000 participants for screening from the employer companies. Screening participants are invited to answer a wellbeing questionnaire (Aava Virta questionnaire, Work Ability Index questionnaire) and give blood samples and physiological measurements, including weight, height, waist circumference, neck circumference and blood pressure. All subjects participating in screening will receive the results from wellbeing questionnaire immediately and they receive the results from blood test within few weeks.

Of these 2000 screened persons, a total of 300 high-risk (according to ApoB/ApoA1) individuals and 600 medium-risk individuals will be selected to participate in the coaching phase. These participants are randomly split into treatment and control groups, so that eventually 150 high-risk and 300 medium-risk individuals are placed in both groups. Therefore, a total of 900 subjects carry forward to the coaching phase and in 1100 subjects the study ends.

All 900 subjects entering coaching phase receive home a Firstbeat Bodyguard 2 device with instructions for performing Firstbeat wellbeing analysis. After the measurement the device is posted back for analysis according to instructions. The results and feedback from this test is received in the end of the study after the coaching phase.

Stage 2: Coaching phase Within the coaching groups, participants in the high-risk category and treatment group undergo an individual coaching program. Participants in the medium-risk category undergo a group coaching program with similar aims. Both coaching programs last 10 weeks during which there are 8 almost weekly coaching sessions at the subjects worksite or near vicinity. Both coaching programs aim in reducing cardiometabolic risk factors and improving subjective well-being. The topics of the lifestyle coaching are 1) nutrition, 2) physical activity, 3) sleep and stress and 4) the long-term maintenance of lifestyle changes. The aims and methods in each coaching topic is based on Finnish recommendations on the topic. The coaching sessions include mostly discussions but in the sessions focusing more on physical activity there are also sessions including activity.

In the halfway (5 weeks) of coaching phase, a second blood sampling and Aava wellbeing questionnaire are taken from all subjects (both coaching and control groups). In the end of the coaching phase (10 weeks) blood samples, Aava wellbeing questionnaire, Work Ability Index -questionnaire and physiological measurements are taken the last time. At this stage a second Firstbeat analysis is also performed. BBI-15 questionnaire is administered before and after the coaching phase. An open ended questionnaire regarding lifestyle change motivators and experiences before, during and after the coaching phase is administered to all participants. Also, a small subset (20 persons) of subjects takes in interviews to delve more detailed to the experiences during the study.

End of coaching phase and study - start of feedback and analysis After the coaching phase has ended and the subjects (coaching and their control groups) have received all the results (wellbeing questionnaire, blood tests and Firstbeat results) for the study and feedback sessions will be held for all. Willing subjects also receive the results from the gene test in form of PRS scores ie. total genetic risk for three areas of health: heart disease, type 2 diabetes and obesity. THL gene results do not identify single gene variants. After this feedback session the study has ended for the subject.

After all data in the study has been gathered starts the analysing and reporting phase for the researchers. At this stage the researchers can retrieve data from Aava patient records to analyse the effect of earlier diagnoses and findings. The information retrieved relate to ICD-10 diagnosis codes C00-C97 (malignant neoplasms), E00-E89 (endocrine, nutritional and metabolic diseases), F00-F99 (mental, behavioral and neurodevelopmental disorders), I00-I99 (diseases of the circulatory system) and M00-M99 (diseases of the musculoskeletal system and connective tissue) as these diagnostic codes can be important background factors for biomarkers of CVD and Type 2 diabetes risk and to some of the secondary endpoints like workability.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Age 18 - 65 years
3. Male or female with at least 1/3 of each gender
4. Adequate Finnish or English* skill to comprehend study-related instructions and questionnaires

Exclusion Criteria:

1. Suspected high probability to travel for more than one working day a week during the trial period according to the investigator's assessment
2. History of a major cardiovascular event (myocardial infarction, coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), stroke, or transient ischemic attack) within the previous 6 months
3. Diagnosed type 1 or type 2 diabetes requiring treatment
4. History of malignant disease such as cancer within five years prior to recruitment
5. Lipid-lowering medication (such as any statin or ezetimibe) or medication for obesity (such as orlistat or liraglutide)
6. Pregnancy
7. Use of cardiac pacemaker or history of atrial fibrillation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
ApoB/ApoA1 | 10 weeks
  Ratio of ApoB to ApoA1 concentration
hs-CRP | 10 weeks
  Measure of low-grade inflammation
TG | 10 weeks
  Fasting triglyceride levels
Fasting blood glucose | 10 weeks
  Fasting blood glucose

SECONDARY OUTCOMES:
Workability | 10 weeks
  Workability assessed by Work Ability Index
Work disability | 10 weeks
  Workability assessed by Work Disablity Prediction Score
Blood pressure, both systolic and diastolic | 10 weeks
  Blood pressure, both systolic and diastolic
Waist circumference | 10 weeks
  Waist circumference
Heart Rate Variability | 10 weeks
  Heart rate variability measurement
Virta Index | 10 weeks
  Self reported data in Virta Index

CONTACTS AND LOCATIONS:
Overall Officials: Eira Roos, PhD, Principal Investigator — Aava Medical
Locations (1):
- Aava Medical, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Shiri R, Vaananen A, Mattila-Holappa P, Kauppi K, Borg P. The Effect of Healthy Lifestyle Changes on Work Ability and Mental Health Symptoms: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Oct 13;19(20):13206. doi: 10.3390/ijerph192013206. PMID 36293787

DOCUMENTS (1):
  • Informed Consent Form (2020-03-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT04633876/ICF_000.pdf